CLINICAL TRIAL: NCT00806936
Title: A 16-week Multicentre, Open Label, Non-interventional, Observational Study to Investigate the Status of Human Insulin or Insulin Analogue Treatments With Focusing on Efficacy and Safety in Type 2 Diabetes Subjects Inadequately Controlled With Two or More Oral Antidiabetic Drugs in China
Brief Title: Observational Study to Investigate the Efficacy and Safety of Human Insulin or Insulin Analogue Treatments in Type 2 Diabetes Subjects
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3675
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A
  Interventions: Drug: human insulin
- B
  Interventions: Drug: insulin analogue

INTERVENTIONS:
Drug: human insulin — Any kind of human insulin administered at the discretion of the physician
  Groups: A
Drug: insulin analogue — Any kind of insulin analogue administered at the discretion of the physician
  Groups: B

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to investigate the percentage of patients reaching the treatment target on blood glucose control after treatment with either human insulin or insulin analogues in type 2 diabetes subjects inadequately controlled with two or more oral antidiabetic drugs in China. Further the safety profiles will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* After the investigator has taken the decision to use human insulin or insulin analogues to treat the subject, any type 2 diabetic previously inadequately controlled with two or more OADs is eligible for the study
* The selection of the subjects will be at the discretion of the individual investigator

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Subjects who are unlikely to comply with protocol requirements, e.g. uncooperative attitude, inability to return for the final visit
* Subjects who previously enrolled in this study
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* The receipt of any investigational product within 3 months prior to this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetic subjects inadequately controlled with two or more oral antidiabetic drugs (OAD) and currently treated with either human insulin or insulin analogues at the discretion of physicians
Sampling Method: Non-Probability Sample
Enrollment: 4847 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving HbA1c below 7.0% | at 16 weeks

SECONDARY OUTCOMES:
HbA1c change from baseline | at 16 weeks
Incidence of major, minor and symptoms only hypoglycaemic episodes | at 16 weeks
Comparison of scores of Insulin Treatment Appraisal Scale (ITAS) | at baseline and at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com